CLINICAL TRIAL: NCT05592197
Title: Safety and Efficacy of External Beam Radiation Plus Transarterial Chemoembolization and Lenvatinib vs Transarterial Chemoembolization and Lenvatinib in Advanced Hepatocellular Carcinoma With Portal Vein Tumor Thrombus
Brief Title: Safety and Efficacy of Radiation Plus TACE and Lenvatinib in Advanced HCC With PVTT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This is a sub-study of another one.
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming Kuang, Professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HCC202211
Record Dates: First submitted 2022-10-20; First posted 2022-10-24 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Advanced Hepatocellular Carcinoma
MeSH Terms: interventions — lenvatinib

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RT+TACE+Lenvatinib (Experimental): Patients in RT+TACE+Lenvatinib group will take oral lenvatinib first and receive TACE one day after oral administration of lenvatinib. RT will begin within 4 weeks after the first TACE.
  Interventions: Drug: Lenvatinib; Procedure: TACE; Radiation: External beam radiation (RT)
- TACE+Lenvatinib (Active Comparator): Patients in TACE+Lenvatinib group will take oral lenvatinib first and receive TACE one day after oral administration of lenvatinib.
  Interventions: Drug: Lenvatinib; Procedure: TACE

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib will be initially provided to patients first (dose: 8 mg qd for patients < 60 kg, and 12 mg qd for patients ≥ 60 kg)
Procedure: TACE — TACE will be performed one day after oral administration of lenvatinib. Either cTACE or DEB-TACE can be used, depending on the condition of each center.
Radiation: External beam radiation (RT) — RT will be given within 4 weeks after the first TACE with linear accelerator-based photon beams. Gross tumor volume is defined as intrahepatic tumor and vascular invasion including a 1-cm margin into the contiguous HCC. Prescription dose will be 4500-6000 cGy in 25 fractions.
  Arms: RT+TACE+Lenvatinib

SUMMARY:
This is a multicentri prospective cohort study to investigate the safety and efficacy of external beam radiation (RT) combined with transarterial chemoembolization (TACE) and lenvatinib vs TACE and lenvatinib in the treatment of advanced hepatocellular carcinoma (HCC) with portal vein tumor thrombus (PVTT).

ELIGIBILITY:
Inclusion Criteria:

1. age 18-75 years;
2. histologically or cytologically or clinically confirmed diagnosis of HCC;
3. presenting with PVTT and at least one measurable intrahepatic lesion on the basis of modified Response Evaluation Criteria in Solid Tumors (mRECIST); an intrahepatic lesion consisting of a single tumor (≤ 10.0 cm) or multiple tumors (≤ 3 foci) with the tumor burden < 50%;
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1;
5. Child-Pugh class A or B;
6. life expectancy of at least 3 months;
7. satisfactory blood, liver, and kidney function parameters. The acceptable blood, liver, and kidney parameters were (1) neutrophil count ≥ 1.5 × 109/L; (2) platelet count ≥ 60 × 109/L; (3) hemoglobin concentration ≥ 90 g/L; (4) serum albumin concentration ≥ 30 g/L; (5) bilirubin ≤ 50 μmol/L; (6) AST and ALT < 5 × upper limit of normal (ULN) and alkaline phosphatase < 4 × ULN; (7) extended prothrombin time < 6 seconds of ULN; and (8) serum creatinine < 1.5 × ULN.

Exclusion Criteria:

1. history of liver and adjacent tissue radiation;
2. medical history of hepatic decompensation, such as hepatic encephalopathy and esophageal or gastric variceal bleeding;
3. extrahepatic spread;
4. combination with other malignant diseases;
5. contraindications for TACE;
6. pregnant and lactating women;
7. severe dysfunction of the heart, kidney, or other organs;
8. hypersensitivity to intravenous contrast agents;
9. with HIV, syphilis infection;
10. allogeneic organ transplant recipients;
11. suffering from mental and psychological diseases may affect informed consent;
12. unable to take oral medication;
13. active gastric or duodenal ulcers within 3 months before enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to 2 years
  OS is defined as the time from the first day of lenvatinib oral administration to death, regardless of disease recurrence.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 2 years
  PFS is defined as the time from the first day of lenvatinib oral administration to progression or death.
Objective Response Rate (ORR) | Up to 2 years
  ORR is defined as the percentage of patients who have achieved complete response (CR) or partial response (PR), as measured by modified Response Evaluation Criteria in Solid Tumors (mRECIST) criteria.
Disease Control Rate (DCR) | Up to 2 years
  DCR is defined as the percentage of patients who have achieved CR, PR or stable disease(SD), as measured by mRECIST criteria.
ncidence of Adverse Events (AE) | Up to 2 years
  The percentage of patients who suffer adverse events from the first day of lenvatinib oral administration to last follow-up, assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Kuang, Ph.D., Study Chair — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peng Z, Fan W, Zhu B, Wang G, Sun J, Xiao C, Huang F, Tang R, Cheng Y, Huang Z, Liang Y, Fan H, Qiao L, Li F, Zhuang W, Peng B, Wang J, Li J, Kuang M. Lenvatinib Combined With Transarterial Chemoembolization as First-Line Treatment for Advanced Hepatocellular Carcinoma: A Phase III, Randomized Clinical Trial (LAUNCH). J Clin Oncol. 2023 Jan 1;41(1):117-127. doi: 10.1200/JCO.22.00392. Epub 2022 Aug 3. PMID 35921605
- [Background] Abulimiti M, Li Z, Wang H, Apiziaji P, Abulimiti Y, Tan Y. Combination Intensity-Modulated Radiotherapy and Sorafenib Improves Outcomes in Hepatocellular Carcinoma with Portal Vein Tumor Thrombosis. J Oncol. 2021 Dec 3;2021:9943683. doi: 10.1155/2021/9943683. eCollection 2021. PMID 34899910
- [Background] Yoon SM, Ryoo BY, Lee SJ, Kim JH, Shin JH, An JH, Lee HC, Lim YS. Efficacy and Safety of Transarterial Chemoembolization Plus External Beam Radiotherapy vs Sorafenib in Hepatocellular Carcinoma With Macroscopic Vascular Invasion: A Randomized Clinical Trial. JAMA Oncol. 2018 May 1;4(5):661-669. doi: 10.1001/jamaoncol.2017.5847. PMID 29543938